CLINICAL TRIAL: NCT07309471
Title: Pharmacokinetics of Didehydro-LSD (DDH-LSD) Compared With LSD
Acronym: DDH-LSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2023-01737;am23Liechti3
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: LSD Reaction
Keywords: DDH-LSD; LSD; Psychedelics; Psychoactive substances; Pharmacokinetics; Pharmacodynamics; Healthy volunteers; 5-HT2A agonist
MeSH Terms: interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: Part 1: Open lable, within-subject, dose-escalation study of DDH-LSD to identify a dose producing measurable psychoactive effects.
  Part 2: randomized, double-blind, placebo-controlled, balanced cross-over study comparing DDH-LSD with LSD and placebo, allowing direct assessment of pharmacokinetics, duration of action, and subjective effects. Each participant completes multiple supervised study sessions separated by washout periods.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DDH-LSD (Experimental): Participants receive a single dose of DDH-LSD at the dose determined in Substudy 1. The session lasts approximately 13 hours with monitoring of subjective, physiological, and pharmacokinetic effects.
  Interventions: Drug: DDH-LSD
- LSD (Active Comparator): Participants receive a single 0.1 mg dose of LSD. The session lasts approximately 13 hours with monitoring of subjective, physiological, and pharmacokinetic effects.
  Interventions: Drug: LSD
- Placebo (Placebo Comparator): Participants receive a placebo dose. The session lasts approximately 13 hours with monitoring of the same parameters to control for expectancy and procedural effects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DDH-LSD — Single oral dose of DDH-LSD at the dose determined in Substudy 1. Participants are monitored for 13 hours for pharmacokinetics, subjective effects, autonomic responses, and safety parameters.
  Arms: DDH-LSD
Drug: LSD — Single oral dose of 0.1 mg LSD. Participants are monitored for 13 hours for pharmacokinetics, subjective effects, autonomic responses, and safety parameters.
  Arms: LSD
Drug: Placebo — Single oral administration of placebo. Participants are monitored for 13 hours under identical conditions to control for expectancy and procedural effects.
  Arms: Placebo

SUMMARY:
This study investigates DDH-LSD, a novel LSD-like compound expected to have a shorter duration of action than LSD. In healthy volunteers, pharmacokinetics, safety, and subjective effects, will be assessed and compare with LSD in a controlled cross-over study.

DETAILED DESCRIPTION:
LSD is a classical serotonergic psychedelic that produces profound alterations in perception and consciousness, primarily through 5-HT2A receptor agonism. Numerous LSD analogs have emerged in recent years, some functioning as prodrugs of LSD, while others show distinct pharmacological characteristics. DDH-LSD is a newly synthesized lysergamide with LSD-like receptor activity but faster metabolism in vitro, suggesting a shorter elimination half-life and potentially briefer psychedelic effects.

This study consists of two parts.

Substudy 1 is an open-label dose-escalation trial in which healthy participants receive increasing doses of DDH-LSD to identify a dose that produces clear but tolerable psychoactive effects.

Substudy 2 is a randomized, double-blind, placebo-controlled cross-over study comparing the selected DDH-LSD dose with LSD and placebo. Each participant completes multiple supervised study days with comprehensive assessment of subjective effects, physiological responses, and pharmacokinetics.

The goal is to provide first-in-human data on DDH-LSD, characterize its effect profile, and evaluate how its duration of action compares with LSD.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years old
2. Sufficient understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study
6. Abstaining from xanthine-based liquids from the evenings prior to the study sessions and during the sessions
7. Willing not to operate heavy machinery within 48 h of substance administration
8. Willing to use effective contraceptive measures throughout study participation
9. Body mass index between 18-32 kg/m2

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Use of hallucinogenic substances (not including cannabis) more than 20 times or any time within the previous two months
6. Pregnancy or currently breastfeeding
7. Participation in another clinical trial (currently or within the last 30 days)
8. Use of medication that may interfere with the effects of the study medication
9. Tobacco smoking (>10 cigarettes/day)
10. Consumption of alcoholic beverages (>20 drinks/week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Determine effective DDH-LSD dose | During each 13-hour study session.
  Identify the dose of DDH-LSD that produces clear psychoactive effects.
Compare duration of action and elimination half-life | During each 13-hour study session.
  Compare DDH-LSD with LSD and placebo regarding elimination half-life and duration of subjective effects.

SECONDARY OUTCOMES:
Pharmacokinetics of DDH-LSD | During each 13-hour study session
  Measure plasma concentration over time
Subjective effects: Visual Analog Scales (VAS) | During each 13-hour study session
  Assess subjective alterations in consciousness using 100 mm horizontal lines (0 = "not at all", 100 = "extremely"). Multiple items (e.g., "any drug effect", "good drug effect", "high", "anxiety") are administered repeatedly during sessions to capture intensity and time course of drug effects.
Subjective effects: Adjective Mood Rating Scale (AMRS / EWL60S) | Following each 13-hour study session
  A 60-item Likert scale assessing six dimensions of mood (activation, positive mood, extraversion, introversion, inactivation, emotional excitability). Scores range from 0-100 per subscale, with higher values indicating greater intensity of the dimension.
Subjective effects: 5-Dimensions of Altered States of Consciousness (5D-ASC) | Following each 13-hour study session
  A 94-item questionnaire assessing altered consciousness, perception, mood, and derealization/depersonalization. Scores 0-100 per subscale, with higher values indicating stronger alteration of consciousness.
Subjective effects: Spiritual Realm Questionnaire (SRQ) | Following each 13-hour study session
  A 65-item visual rating scale assessing spiritual and psychedelic experiences across four dimensions (spirituality, human condition, personal problem solving, worldview/beliefs). Scores 0-100 per subscale, higher values indicate stronger experience.
Subjective effects: States of Consciousness Questionnaire (SCQ / MEQ) | Following each 13-hour study session
  A 100-item questionnaire with a 43-item Mystical Experience Questionnaire (MEQ) embedded. Scores 0-100% per domain, with higher percentages reflecting stronger mystical-type experiences.
Effect on heart rate (HR) | During each 13-hour study session
Effect on blood pressure | During each 13-hour study session
Effect on body temperature | During each 13-hour study session
Subjective effects: Scale of Positive and Negative Experience (SPANE) | Before each 13-hour study session
  A 12-item questionnaire measuring positive and negative affect. Subscales range 0-24, with higher scores indicating greater positive or negative affect; the overall balance score reflects general well-being.
Subjective effects: Psychological Insight Questionnaire (PIQ) | Following each 13-hour study session
  A 14-item questionnaire assessing insight into emotions, behavior, beliefs, or relationships. Items rated 0-5 (0 = "not at all", 5 = "extremely"), higher scores indicate greater perceived psychological insight.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Liechti, Prof.MD, Study Chair — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland